CLINICAL TRIAL: NCT02234388
Title: Undifferentiated Connective Tissue Disease Registry
Acronym: UCTD Registry
Status: Recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-311; Robin J. Sillau Fund (Other Grant/Funding Number: Robin J. Sillau Fund for Connective Tissue Disease Research)
Record Dates: First submitted 2014-09-03; First posted 2014-09-09 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Undifferentiated Connective Tissue Disease
Keywords: connective tissue disease; registry; hospital for special surgery
MeSH Terms: conditions — Undifferentiated Connective Tissue Diseases; Connective Tissue Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Registry Participants: All patients who participate in the UCTD Registry will be put into this cohort and observed over approximately 3 years.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — There are no interventions associated with this registry as it is purely observational.

SUMMARY:
This registry has been established to gain a better understanding of the clinical and emotional presentations of patients with undifferentiated connective tissue disease.

DETAILED DESCRIPTION:
The purpose of this research registry is to gather information about clinical symptoms and laboratory test results in patients with undifferentiated connective tissue disease (UCTD). Analysis of this information may help to better predict the prognosis for patients with this form of autoimmune disease, and may identify risk factors for progression to more specific connective tissue diseases such as systemic lupus. This is done by collecting information from your medical records including clinical history, physical examination, and lab test results, and by asking you questions about specific symptoms you may have such as joint pain, rashes, and other common symptoms of UCTD. This information will be stored in a database, and used at a later time for research studies. All future research studies using information in this registry will be subject to oversight by HSS's Institutional Review Board (which is responsible for oversight of research at HSS involving human subjects). All patients who seek or receive medical care at HSS for undifferentiated connective tissue disease will be invited to participate in this registry.

Most future research studies involving this registry will only use the information in this registry, and therefore will not require the further involvement or additional informed consent of participants in the registry. But the information in this registry may also be used to identify patients who may be eligible to participate in certain future research studies conducted by HSS that relate to their particular disease, condition, or treatment and for which information is needed that is not in the registry. If you are identified (based on information about you in the registry) as being potentially eligible for a future research study that relates to your particular disease, condition, or treatment, you may be contacted to find out if you would be interested in participating in the research study. If you are interested, the research study would be fully explained to you, and you would have to give your informed consent before you could participate. If you participate in this registry, you will not be required to participate in any future research study that HSS contacts you about.

By participating in this registry, you will not be asked to do anything that would not ordinarily be done as a matter of routine care at HSS including clinical assessments, laboratory tests and radiology procedures. During your routine visits we will be recording all of the information about you that relates to your disease, condition, or treatment and will include that information in the registry. Your participation will involve a minimum of one yearly visit at the time of your visit to your own rheumatologist. Most study visits are expected to last 10 - 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Any patient under the care of an HSS rheumatologist
* Positive ANA or a positive anti-ds DNA, anti-Ro/SS-A or other autoantibody on 2 or more occasions at least 12 weeks apart
* One or more signs or symptoms of connective tissue disease, including but not limited to arthralgia, arthritis, myalgia, rash, sicca symptoms, pericarditis, pleuritis, pulmonary symptoms, peripheral neuropathy, photosensitivity, alopecia, oral or nasal ulcers, leucopenia, anemia, and abnormal nailfold capillaroscopy

Exclusion Criteria:

* Patients who meet criteria for well defined CTD including SLE, rheumatoid arthritis, polymyositis or dermatomyositis, systemic sclerosis, or antiphospholipid syndrome
* Patients who are less than 18
* Those unable to give informed consent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under the care of any HSS rheumatologist that have been diagnosed with undifferentiated connective tissue disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-03; Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in SF-36 Score | 3 years
  Patient questionnaire that measures health-related quality of life.
Change in Fatigue Severity Scale Score | 3 years
  Evaluates the impact of fatigue on the patient.
Change in Beck Depression Inventory Score | 3 years
  Self-reported depression severity questionnaire
Connective Tissue Disease Criteria | 3 years
  The physician will monitor which characteristics from each connective tissue disease the patient presents with. This will show how UCTD progresses and what the most prominent characteristics of the disease are.

SECONDARY OUTCOMES:
CBC | 3 years
  Patients may have this clinical lab test ordered to monitor their hemoglobin, hematocrit, and platlet counts.
Comprehensive Metabolic Panel | 3 years
  Patients may have this clinical laboratory test ordered to monitor their electrolytes, creatinine, glucose levels, phosphates, and blood protein levels.
Cholesterol Profile | 3 years
  Patients may have this clinical laboratory test ordered to monitor their blood cholesterol levels.
Urinalysis | 3 years
  Patients may have this clinical laboratory test ordered to monitor their health and the presence of any infections.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States